CLINICAL TRIAL: NCT06458491
Title: Evolution of Urinary Symptoms After Use of TENSI+ Posterior Tibial Nerve Stimulation for Overactive Bladder
Brief Title: Urinary Symptoms After Posterior Tibial Nerve Stimulation
Acronym: TENSI
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0590
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Posterior Tibial Nerve Stmulation
Keywords: overactive bladder; Posterior Tibial Nerve Stmulation
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TENSI+ posterior tibial nerve stimulation for overactive bladder: patients who have benefited from treatment with the TENSI+ device in the context of overactive bladder
  Interventions: Device: Evolution of urinary symptoms

INTERVENTIONS:
Device: Evolution of urinary symptoms — Evolution of urinary symptoms 3 months after the start of use of the TENSI+ device

SUMMARY:
Overactive bladder (OAB) is a common syndrome affecting 7 million people in France, very often of idiopathic origin.

Current therapeutic management of OAB primarily involves hygiene and diet rules, patient education, behavioral measures with bladder reprogramming or even perineo-sphincter rehabilitation. However, the modalities of this conservative non-drug treatment are poorly defined and there is uncertainty as to their effectiveness.

In the event of persistent symptoms, the management of OAB is essentially based on the prescription of an anticholinergic medication. The effectiveness of anticholinergics has been established through numerous randomized clinical trials and meta-analyses. But the side effects of anticholinergics are known and some are very common (particularly dry mouth and constipation).

The principle of the posterior tibial nerve stimulation (TNS) by implanted (percutaneous) or adhesive (transcutaneous) electrode is to stimulate the sensory afferent pathways and to ensure negative feedback on the bladder. Posterior tibial nerve stimulation is a non-invasive therapeutic alternative that has demonstrated its effectiveness through numerous clinical studies mainly using a device for percutaneous use with a weekly stimulation session.

TNS is also possible transcutaneously (TENS) with daily 20-minute stimulation of the ankle, in the form of a self-administered treatment at home, over a period of 3 months. This treatment modality seems equivalent to the percutaneous approach.

Given its numerous advantages, the use of TENS is therefore expanding, and is currently recommended by many learned societies (SIFUD, AFU).

In this study, we wish to evaluate the TENSI+ medical device which uses transcutaneous posterior tibial nerve stimulation and which is offered in routine practice to patients with idiopathic or neurological overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* women over 18
* patients who have benefited from treatment with the TENSI+ device in the context of overactive bladder
* intervention between April 2023 and February 2024
* person having expressed his non-opposition

Exclusion Criteria:

* inability to understand the information given
* person deprived of liberty
* person under guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This study concerns all patients who have benefited from treatment with the TENSI+ device in the context of overactive bladder between April 2023 and February 2024.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Evolution of urinary symptoms | 3 months after the start of treatment
  change in the "overactive bladder" score obtained by the USP questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Department of obstetrics, Femme Mère Enfant Hospital, Lyon, France, Bron, France